CLINICAL TRIAL: NCT03733535
Title: A Mechanistic Pilot Open-label Study to Evaluate the Effect of Benralizumab on Airway Function and Inflammation in Patients With Severe, Poorly-controlled Eosinophilic Asthma Using Inhaled Hyperpolarized 129-Xenon MRI
Brief Title: Evaluating the Effect of Benralizumab in Severe, Poorly-controlled Eosinophilic Asthma Using Inhaled Hyperpolarized 129-Xenon MRI
Acronym: AERFLO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Grace Parraga (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROB0042
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Eosinophilic
Keywords: Benralizumab; Xenon
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Open-label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Benralizumab 30mg subcutaneous injection on study days 0, 28 and 56 and 1.0 L 129-Xenon/4-Helium mixture, twice per visit, on days 0, 14, 28 and 112.
  Interventions: Drug: Benralizumab; Drug: 129 Xenon

INTERVENTIONS:
Drug: Benralizumab — Benralizumab is an interleukin-5 receptor alpha-directed cytolytic monoclonal antibody
  Other Names: Fasenra
Drug: 129 Xenon — 1.0 L of 129-Xenon/4-Helium mixture to acquire MRI images
  Other Names: 129-Xe

SUMMARY:
The purpose of this study is to evaluate the effect of a drug called benralizumab in individuals with severe, poorly controlled asthma with eosinophilic airway inflammation. Eosinophils are a type of white blood cell that help fight off infections. Some people with asthma have too many eosinophils in their airways and blood, which can cause airway inflammation. Benralizumab is a new drug that is Health Canada approved and has been shown to rapidly eliminate eosinophils. It has been used in patients with severe asthma to improve lung function and reduce flair-ups, also known as exacerbations. Magnetic Resonance Imaging (MRI) is an imaging tool that can look at the structure of the lungs when a subject inhales a xenon gas mixture. In healthy individuals, the gas fills the lungs evenly, but in individuals with lung disease, some of the areas of the lungs are not filled by the gas and the image looks patchy. These patchy areas are called ventilation defects and they contribute to reduced lung function. The goal of the study is to see if treatment with benralizumab will improve these ventilation defects, overall lung function and blood and sputum eosinophil levels. Subjects will receive treatment with benralizumab a total of 3 times, 4 weeks apart. Before and after treatment, subjects will undergo a series of MRI tests, breathing tests, blood and sputum analysis and a series of questionnaires to evaluate daily quality of life. The hypothesis is that ventilation defects will significantly improve after benralizumab treatment, and that this improvement will be different based on how long the patient has had asthma.

DETAILED DESCRIPTION:
This is an open-label, single arm, pilot study in patients with severe, poorly-controlled eosinophilic asthma to quantify hyperpolarized 129-Xenon MRI ventilation defect percent (VDP) before and after benralizumab therapy administered every 4 weeks for the first three injections (subcutaneous injection). Male and female patients between 18 and 70 years of age will be screened (Enrolment, Visit 1) and those that satisfy all inclusion and exclusion criteria will undergo five additional two-hour study visits (Visit 2=Day 0/baseline, Visit 3=Day 14±2 days and Visit 4=Day 28±2 days, Visit 5=Day 56±2 days, Visit 6=112±2 days) which will involve spirometry, plethysmography for airways resistance (Raw) and lung volumes, forced oscillation technique (FOT), multiple breath nitrogen washout (MBNW) for the lung clearance index (LCI) and 129-Xenon MRI pre- and post-bronchodilator, with the exception of Visit 5, which will not include MRIs. At all visits fractional exhaled nitric oxide (FeNO) will be measured pre-bronchodilator. The Asthma Control Questionnaire (ACQ-6), the Asthma Quality of Life Questionnaire (AQLQ) and the St. George's Respiratory Questionnaire (SQRQ) will be completed at all visits except Visit 3. Sputum induction will be performed on Visits 2 and 4 to measure sputum eosinophils, and blood samples will be performed on Visits 1 and 4 to measure blood eosinophils. Participants that satisfy all inclusion and exclusion criteria will complete a total of six study visits. Upon study enrolment, all participants will be allocated to a benralizumab treatment arm (30 mg injection after completion of study assessments on Visit 2/Day 0, Visit 4/Day 28 and Visit 5/Day 56). After Visit 6/Day 112, all participants will be offered participation in the AstraZeneca Patient Support Program to receive benralizumab therapy on Day 112 and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands study procedures and is willing to participate in the study as indicated by the patient's signature
* Provision of written, informed consent prior to any study specific procedures
* Males and females with a clinical diagnosis of asthma aged 18 to 70 years, inclusively, at the time of Visit 1 (enrolment), under the care of a respirologist
* Patient is a current non-smoker, having not smoked tobacco or cannabis for at least 12 months prior to the study with a tobacco smoking history of no more than 1 pack-year (i.e., 1 pack per day for 1 year)
* Women of childbearing potential (after menarche) must use a highly effective form of birth control (confirmed by the investigator or designee). A highly effective form of birth control includes true sexual abstinence, a vasectomized sexual partner, Implanon®, female sterilization by tubal occlusion, any effective intrauterine device (IUD)/levonorgestrel intrauterine system (IUS), Depo-Provera (trademark) injections, oral contraceptive and Erva Patch (trademark) or Nuvaring (trademark)
* Women of childbearing potential (after menarche) must agree to use a highly effective form of birth control, as defined above, from enrolment, throughout the study duration, and within 16 weeks after last dose of study drug, and have negative serum pregnancy test result on enrolment
* Male patients who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of the study drug until 16 weeks after last dose
* Patient has documented treatment with medium- to high-dosage inhaled corticosteroids (ICS) (>250μg fluticasone dry powder formulation equivalents total daily dosage) and a long-acting β2-agonist (LABA) for at least 12 months prior to enrolment.
* Patient has been treated with high dose ICS (at least 500μg/day fluticasone propionate dry powder formulation or equivalent daily) and LABA for at least 3 months prior to Visit 2 with or without oral corticosteroids (OCS) and additional asthma controllers
* Patient demonstrates pre-bronchodilator (Pre-BD) forced expiratory volume in one second ˂ 80% predicted
* Patient demonstrated significant bronchodilator reversibility (≥ 12% AND ≥ 200 mL improvement) or positive methacholine challenge test (PC20 < 4.0 mg/ml) in past 24 months
* Patient has blood eosinophils ≥ 300 cells/μl
* Patient has ACQ-6 ≥ 1.5 at visit 1
* Patient has a history of poorly controlled asthma

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand written material
* Patient has clinically important pulmonary disease other than asthma (e.g. active lung infection, chronic obstructive pulmonary disease, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha-1 antitrypsin deficiency and primary ciliary dyskinesia) or been diagnosed with pulmonary or systemic disease other than asthma that is associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome), except for those atopic conditions that can be associated with asthma (e.g. allergic rhinitis, sinusitis with or without polyposis, eczema, and eosinophilic esophagitis)
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Qualified Investigator and/or could affect the safety of the patient throughout the study, influence the findings of the study or their interpretations, or impede the patient's ability to complete the entire duration of the study, as assessed by the Qualified Investigator.
* Known history of allergy or reaction to the study drug formulation
* History of anaphylaxis to any biologic therapy
* A helminthic parasitic infection diagnosed within 24 weeks prior to the date of informed consent that has not been treated with or failed to respond to standard-of-care therapy
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date of informed consent
* Use of immunosuppressive medication (including but not limited to methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid or any experimental anti-inflammatory therapy) within 3 months prior to the date of informed consent
* Chronic maintenance prednisone for the treatment of asthma is allowed
* Clinically significant asthma exacerbation, in the opinion of the investigator, including those requiring the use of OCS, or an increase in maintenance dosage of OCS 14 days prior to the date of informed consent
* Receipt of immunoglobulin or blood products within 30 days prior to the date of informed consent
* Receipt of live attenuated vaccines 30 days prior to the date of enrolment
* Receipt of any marketed (e.g., omalizumab) or investigational biologic within 4 months or 5 half-lives prior to the date of informed consent, whichever is longer AND blood eosinophils ≥ 300 cells/µl.
* Receipt of any investigational nonbiologic within 30 days or 5 half-lives prior to enrolment, whichever is longer
* Previously randomized in any benralizumab (MEDI-563) study
* Initiation of new allergen immunotherapy within 30 days prior to the date of informed consent
* Current use of any oral of opthalmic nonselective β-adrenergic antagonist (e.g., propranolol)
* Planned surgical procedure during the conduct of the study
* Concurrent enrolment in another clinical trial
* Patient has donated a unit of blood within 4 weeks prior to Visit 1 or anticipates donating blood at any time during the study
* Patient has history of alcohol or drug abuse within 12 months prior to the date of informed consent
* Patient is a female who is ≤8 weeks post-partum or breast feeding an infant
* Patient is pregnant, or intends to become pregnant during the time course of the study
* Patient is unable to perform MRI breath-hold maneuver
* Patient is unable to perform spirometry maneuver
* Patient is hospitalized or has had a major surgical procedure, major trauma requiring medical attention, or significant illness requiring medical attention within 4 weeks of Visit 1
* Patient has a blood pressure of >150 mmHg systolic or >95 mmHg diastolic on >2 measurements done >5 minutes apart at Visit 1 or Visit 2
* Patient has ECG abnormalities consistent with previous myocardial infarction, hypertrophic cardiomyopathy, ischemic heart disease or conduction system disease
* In the opinion of the investigator, patient suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia
* Patient has implanted mechanically, electrically or magnetically activated device or any metal in their body, which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) - at the discretion of the MRI Technologist.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline airway function measured using 129-Xenon MRI ventilation defect percent | Day 0 and 28
  Changes in VDP

SECONDARY OUTCOMES:
Change from baseline airway function measured using 129-Xenon MRI ventilation defect percent | Day 0, 14 and 112
  Changes in VDP
Change from baseline blood eosinophils | Day 0, 14 and 112
Change from baseline forced expiration volume in one second | Day 0, 14, 28 and 112
  Indicator of pulmonary function
Change from baseline forced vital capacity | Day 0, 14, 28 and 112
  Indicator of pulmonary function
Change from baseline lung volumes | Day 0, 14, 28 and 112
  Indicator of pulmonary function
Change from baseline airways resistance | Day 0, 14, 28 and 112
  Indicator of pulmonary function and inflammation
Change from baseline forced oscillation technique | Day 0, 14, 28 and 112
  Indicator of pulmonary function and inflammation
Change from baseline lung clearance index | Day 0, 14, 28 and 112
  Indicator of pulmonary function
Change from baseline fraction exhaled nitric oxide | Day 0, 14, 28 and 112
  Indicator of pulmonary function and inflammation
Change from baseline in asthma control | Day 0, 28, 56 and 112
  Asthma Control Questionnaire (ACQ-6) is used to evaluate asthma control. The ACQ-6 is scored from 0 to 6, with higher scores indicating more severely uncontrolled asthma.
Change from baseline in asthma-related quality of life | Day 0, 28, 56 and 112
  Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Change from baseline in daily life and perceived well-being | Day 0, 28, 56 and 112
  St. George's Respiratory Questionnaire (SGRQ) evaluates daily life and perceived well-being in relation to asthma and respiratory conditions. The SGRQ is scored from 0-100 with higher scores indicating more limitations.
Change from baseline in Clinician Global Impressions of Change | Day 0 and 112
  The Clinical Global Impressions of Change is an indicator of improvement or decline in clinical status from the perspective of the clinician. It is a scale from 1-7, with lower scores indicating more improvement in clinical status.
Change from baseline in Patient Global Impressions of Change | Day 0 and 112
  The Patient Global Impressions of Change is an indicator of improvement or decline in clinical status from the perspective of the patient. It is a scale from 1-7, with lower scores indicating more improvement in clinical status.

OTHER OUTCOMES:
Explore univariate correlation and linear regression of MRI ventilation defect percent and asthma control as measured by the Asthma Control Questionnaire | Day 112
  The relationship between ventilation defect percent and asthma control, as measured by the Asthma Control Questionnaire (ACQ-6) will be assessed using a univariate correlation analysis and linear regression. The ACQ-6 is scored from 0 to 6, with higher scores indicating more uncontrolled asthma.
Explore univariate correlation and linear regression of MRI ventilation defect percent and asthma-related quality of life as measured by the Asthma Quality of Life Questionnaire | Day 112
  The relationship between ventilation defect percent and asthma-related quality of life as measured by the Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) will be assessed using a univariate correlation analysis and linear regression. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Explore univariate correlation and linear regression of MRI ventilation defect percent and daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire | Day 112
  The relationship between ventilation defect percent and daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire (SGRQ) will be assessed using univariate correlation analysis and linear regression. The SGRQ is scored from 0-100 with higher scores indicating more limitations.
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced expiration volume in one second. | Day 112
  The relationship between ventilation defect percent and forced expiration volume in one second will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced vital capacity | Day 112
  The relationship between ventilation defect percent and forced vital capacity will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and lung volumes | Day 112
  The relationship between ventilation defect percent and lung volumes will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and airways resistance | Day 112
  The relationship between ventilation defect percent and airways resistance will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function, structure and inflammation.
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced oscillation technique | Day 112
  The relationship between ventilation defect percent and forced oscillation technique will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function, structure and inflammation.
Explore univariate correlation and linear regression of MRI ventilation defect percent and lung clearance index | Day 112
  The relationship between ventilation defect percent and lung clearance index will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and sputum measurements of eosinophilia | Day 112
  The relationship between ventilation defect percent and sputum eosinophils will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary structure and sputum eosinophils.
Explore univariate correlation and linear regression of MRI ventilation defect percent and blood measurements of eosinophilia | Day 112
  The relationship between ventilation defect percent and blood eosinophils will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary structure and blood eosinophils.
Explore univariate correlation and linear regression of MRI ventilation defect percent and fraction exhaled nitric oxide | Day 112
  The relationship between ventilation defect percent and airways resistance will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function, structure and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McIntosh MJ, Kooner HK, Eddy RL, Wilson A, Serajeddini H, Bhalla A, Licskai C, Mackenzie CA, Yamashita C, Parraga G. CT Mucus Score and 129Xe MRI Ventilation Defects After 2.5 Years' Anti-IL-5Ralpha in Eosinophilic Asthma. Chest. 2023 Jul;164(1):27-38. doi: 10.1016/j.chest.2023.02.009. Epub 2023 Feb 11. PMID 36781102
- [Derived] McIntosh MJ, Kooner HK, Eddy RL, Jeimy S, Licskai C, Mackenzie CA, Svenningsen S, Nair P, Yamashita C, Parraga G. Asthma Control, Airway Mucus, and 129Xe MRI Ventilation After a Single Benralizumab Dose. Chest. 2022 Sep;162(3):520-533. doi: 10.1016/j.chest.2022.03.003. Epub 2022 Mar 10. PMID 35283104